CLINICAL TRIAL: NCT03122106
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Neoantigen DNA Vaccine Strategy in Pancreatic Cancer Patients Following Surgical Resection and Adjuvant Chemotherapy
Brief Title: Neoantigen DNA Vaccine in Pancreatic Cancer Patients Following Surgical Resection and Adjuvant Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201708105; P50CA196510-01A1 (NIH)
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Cancer of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Personalized neoantigen DNA vaccine (Experimental): * Vaccines will be weeks 1, 5, 9, 13, 17, and 21. Vaccines will occur within +/- 1 week with at least 3 weeks between vaccines. All study injections will be given intramuscularly using TDS-IM system. At each vaccination time point, patients will receive 2 injections of the neoantigen DNA vaccine, 1 injection into each deltoid or lateralis.
  * Minimum observation of 30 minutes. Vital signs will be taken at 30-45 minutes post-immunization. The injection sites will be inspected for evidence of local reaction. Follow up on subject well-being will be performed by telephone on the 1st or 2nd day following each injection. -Post-vaccination follow-up visits are at Week 25 ± 7 days and Week 77 ± 14 days. Additional follow-up visits or telephone contact will be scheduled at Week 129 and annually thereafter if the patient is alive and available for follow-up.
  * At intervals throughout the study (both before and after vaccination) subjects will have blood drawn for immunologic assays.
  Interventions: Biological: Personalized neoantigen DNA vaccine; Device: TDS-IM Electrode Array System; Procedure: Peripheral blood draws

INTERVENTIONS:
Biological: Personalized neoantigen DNA vaccine — -Personalized polyepitope inserts integrating the prioritized neoantigens and mesothelin epitopes will be designed and then synthesized and cloned into the pING parent vector
Device: TDS-IM Electrode Array System — -Ichor Medical Systems
Procedure: Peripheral blood draws — -Enrollment, mid adjuvant chemotherapy, end of chemotherapy, week 1, week 5, week 9, week 13, week 17, week 21, week 25, and week 77

SUMMARY:
This is a phase 1 open-label study to evaluate the safety and immunogenicity of a neoantigen DNA vaccine strategy in pancreatic cancer patients following surgical resection and adjuvant chemotherapy. The neoantigen DNA vaccines will incorporate prioritized neoantigens and personalized mesothelin epitopes and will be administered with an electroporation device. The hypothesis of this study is that neoantigen DNA vaccines will be safe and capable of generating measurable neoantigen-specific CD4 and CD8 T cell responses.

DETAILED DESCRIPTION:
-Subjects will be enrolled within 12 weeks of surgery and standard of care adjuvant chemotherapy will last approximately 12 weeks with an additional 12 weeks of standard of care adjuvant chemotherapy or adjuvant chemoradiation. The first vaccine may be administered following confirmation of disease-free status and within 60 days following date of repeat imaging. From time of enrollment to first vaccine could be up to 45 weeks.

ELIGIBILITY:
A patient will be eligible for the trial only if ALL of the following criteria apply:

Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma; mixed histology will be included as long as the predominant histology is adenocarcinoma.
* Completed an R0 or R1 surgical resection as determined by pathology
* Pathology review demonstrates tumor cellularity no less than 30% in quantities sufficient to obtain 6-8 1mm biopsies from the original FFPE blocks.
* At least 18 years of age.
* Life expectancy of > 12 months.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * white blood cells (WBC) ≥3,000/μL
  * absolute neutrophil count ≥1,500/μL
  * platelets ≥100,000/μL
  * total bilirubin ≤2.5 X institutional upper limit of normal (ULN)
  * AST/ALT≤ 2.5 X institutional upper limit of normal
  * creatinine ≤1.5 X institutional upper limit of normal
* International Normalized Ratio (INR) and activated partial thromboplastin time (PTT) < 1.5 x ULN provided the patient is not on anticoagulation therapy.
* Patients who have had a stent placed for biliary obstruction can be included in the study provided serum bilirubin at time of enrollment is within protocol limits.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.

Patients may be consented prior to receiving adjuvant therapy, or during the course of adjuvant therapy. Adjuvant therapy must meet the following criteria below for enrollment to the trial:

* Initiation of adjuvant chemotherapy within 12 weeks of surgery
* Completion of at least 4 months of adjuvant chemotherapy with gemcitabine/capecitabine or similar adjuvant chemotherapy at the discretion of the patient's medical oncologist.
* Additional chemoradiation therapy as recommended by the patient's medical oncologist.
* Reimaging within 4 weeks of last dose of chemotherapy demonstrates no evidence of recurrent disease and CA 19-9 is less than 92.5 u/mL
* Dose modifications and/or delays in adjuvant chemotherapy is at the discretion of the treating physician -There is a 1 week washout prior to Day 1 of vaccine for patients on daily systemic steroids at doses exceeding 10 mg prednisone.

Exclusion Criteria:

* Evidence of neuroendocrine tumor, duodenal adenocarcinoma, or ampullary adenocarcinoma.
* Received neoadjuvant chemotherapy for their pancreatic adenocarcinoma
* Evidence of disease recurrence or metastasis following surgical resection at any time prior to the first vaccination administration. Most patients will undergo restaging midway through adjuvant chemotherapy and at the completion of therapy; however, timing of imaging is at the discretion of the patient's medical oncologist.
* History of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Receiving any other investigational agents, or has received an investigational agent within the last 30 days.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, hepatic renal, and/or other functional abnormality that would jeopardize the health and safety of the participant as determined by the investigator based on medical history, physical examination, laboratory values, and/or diagnostic studies.
* A psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator from the medical history, physical exam, and/or medical record
* History of syncopal or vasovagal episode as determined by medical record and history in the 12 month period prior to first vaccination administration.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right medial deltoid region) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. In the case of asthma or chronic obstructive pulmonary disease taking inhaled corticosteroids that does not require daily systemic corticosteroids is acceptable. Additionally, local acting steroids (topical, inhaled, or intraarticular) will be allowed. Patients on intermittent or short course steroids will be allow if the dose does not exceed 4 mg of dexamethasone (or equivalent) per day for > 7 consecutive days. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant and/or breastfeeding.
* Known HIV-positive status. These patients are ineligible because of the potential inability to generate an immune response to vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2022-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gillanders, M.D., Principal Investigator — Washington University School of Medicine; Daniel Laheru, M.D., Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Personalized Neoantigen DNA Vaccine
Started | 15
Completed | 11
Not Completed | 4
Not completed — Not enough tissue | 1
Not completed — Disease progression during screening | 2
Not completed — Poor RNA quality for vaccine | 1

BASELINE CHARACTERISTICS:
Arm/Group | Personalized Neoantigen DNA Vaccine
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 67 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety of Neoantigen DNA Vaccine as Measured by the Number of Subjects Experiencing Each Type of Treatment-related Adverse Event
Description: * Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0
  * Related indicates possibly, probably, or definitely related to the study treatment
Time Frame: Through week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized Neoantigen DNA Vaccine
Number analyzed (Participants) | 11
Participants
  Abdominal pain | 1
  Bruising | 1
  Chills | 1
  Conjunctivitis | 1
  Fatigue | 2
  Fever | 1
  Injection site pain | 10
  Injection site reaction | 2
  Hypertension | 1
  Muscle soreness | 1
  Myalgia | 10
  Nausea | 1
  Pain | 1

2. Secondary Outcome: Immunogenicity of the Neoantigen DNA Vaccine as Measured by ELISPOT Analysis
Description: Immunogenicity is defined as the number of participants with a neoantigen-specific immune response measured by ELISPOT analysis. A participant is considered a responder if there is a significant increase in the number of neoantigen-specific T cells to at least one neoantigen after vaccination. A significant increase is based on t-test comparing the number of neoantigen-specific T-cells before and after vaccination with p=0.05 for significance.
Time Frame: Through week 77
Population: Participants who are not included in this outcome measure include one who did not have enough tissue, one who had poor quality RNA and a vaccine could not be developed, and 2 who developed disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized Neoantigen DNA Vaccine
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Immunogenicity of the Neoantigen DNA Vaccine as Measured by Multiparametric Flow Cytometry
Time Frame: Through week 77
Population: The multiparametric flow cytometry assay described in the protocol was not sufficiently sensitive to reliably detect neoantigen-specific T cell responses. Additional flow cytometry assays are being performed as an exploratory objective.
Arm/Group | Personalized Neoantigen DNA Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 24 weeks. All-cause mortality was collected from start of treatment through completion of follow-up (estimated to be 73 weeks).
Arm/Group | Personalized Neoantigen DNA Vaccine
All-Cause Mortality (participants affected / at risk) | 5/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Personalized Neoantigen DNA Vaccine (N=11)
Anemia (Blood and lymphatic system disorders) | 3
Iron deficient anemia (Blood and lymphatic system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Injection site pain (General disorders) | 10
Injection site reaction (General disorders) | 2
Pain (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bilateral lower extremity cramping (Musculoskeletal and connective tissue disorders) | 1
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Cold sweats (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT03122106/Prot_SAP_002.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT03122106/ICF_001.pdf